CLINICAL TRIAL: NCT06557317
Title: Examining the Preliminary Efficacy of an In-Person Lifestyle Intervention for Black Female Adolescent/Caregiver Dyads at Risk for Type 2 Diabetes Mellitus
Brief Title: In-Person Lifestyle Program for Black Adolescent Girls at Risk for Type 2 Diabetes
Acronym: BGW In-Person
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0148278
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Behavior, Adolescent; Childhood Obesity; Diabetes Mellitus, Type 2; Pediatric Obesity; Glucose Metabolism Disorders; Metabolic Disease; Endocrine System Diseases; Overweight; Overnutrition; Nutrition Disorders; Body Weight; Diabetes Mellitus
Keywords: Adolescents; In-Person Lifestyle Program; Diabetes prevention; Black girls; Obesity
MeSH Terms: conditions — Adolescent Behavior; Pediatric Obesity; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Overweight; Overnutrition; Nutrition Disorders; Body Weight; Diabetes Mellitus; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Adolescent/Caregiver Dyads (Experimental): Adolescent/Caregiver dyads receive 12-week in-person lifestyle program consisting of a Wellness session, Dance Classes, and an at-home Cooking Experience.
  Interventions: Behavioral: Black Girls for Wellness In-Person

INTERVENTIONS:
Behavioral: Black Girls for Wellness In-Person — Weekly for 12 weeks, adolescent/caregiver dyads will attend 1) an in-person Wellness Session (mindfulness, nutrition lesson, dance class, program reflection) (90 min/wk) and 2) a home cooking experience using ingredients provided at the Wellness Session (60 min/wk).

SUMMARY:
The aim of this study is to look at changes in diabetes-related risk factors in Black adolescent girls who are at risk for type 2 diabetes and their primary female caregiver after both participating in a 12-week in-person lifestyle program.

DETAILED DESCRIPTION:
Enrolled adolescent/caregiver dyads will participate in the 12-week program. Each week, participants will engage in 2 activities: an in-person Wellness Session and an at-home cooking experience using ingredients provided at the Wellness Session.

The study will examine the pre-post difference in overall diet quality, dermal carotenoid levels, physical activity, body composition, and glycemic measures among at-risk black adolescent girls and their caregivers. Investigators hypothesize that after the program, participants' diets will be higher in quality than before.

ELIGIBILITY:
Inclusion Criteria for adolescent participants:

* 12-18 years of age
* self-identify as Black or African American
* have obesity (>=95th percentile BMI)

Exclusion Criteria for adolescent participants:

* pregnant or within 3 months postpartum.
* participated in a formal weight management program within 6 months prior to study.
* currently taking medications or diagnosed with a condition known to influence metabolism, physical activity ability, or cognitive function.
* have previously undergone bariatric surgery.
* have type 2 diabetes.
* unable to speak English or have developmental conditions that interfere with ability to communicate.

Inclusion Criteria for caregiver participants:

* 18 years or older.
* proficiency in speaking English.
* live in the same household as the adolescent who will also be enrolled.
* prepares the majority (>50%) of meals in the household.

Exclusion Criteria for caregiver participants:

* pregnant or within 3 months postpartum.
* unable to speak English or have developmental conditions that interfere with ability to communicate.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Inclusion Criteria for all participants includes biological sex female.
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in diet quality of adolescent participants, as measured by the Healthy Eating Index Scores | Baseline, 12 weeks [end of study]
  Scores are calculated from three 24-hour diet records, range from 0-100. Higher score reflects that higher alignment between one's diet and dietary recommendations from the Dietary Guidelines for Americans.

SECONDARY OUTCOMES:
Change in dermal carotenoids level | Baseline, 12 weeks [end of study]
  Scores are measured using the Veggie Meter device, range from 0-800. Higher score acts as proxy for fruits and vegetables consumption.
Change in percent time sedentary | Baseline, 12 weeks [end of study]
  Accelerometry data will be collected from wrist accelerometers worn by participants for 7 days. Percent time spent on sedentary will be calculated.
Change in percent time spent in light activity | Baseline, 12 weeks [end of study]
  Accelerometry data will be collected from wrist accelerometers worn by participants for 7 days. Percent time spent in light activity will be calculated.
Change in percent time spent in moderate to vigorous activity | Baseline, 12 weeks [end of study]
  Accelerometry data will be collected from wrist accelerometers worn by participants for 7 days. Percent time spent in moderate and vigorous activity will be calculated.
Change in HbA1c | Baseline, 12 weeks [end of study]
  HbA1c will be assessed through a blood draw.
Change in lipid profile | Baseline, 12 weeks [end of study]
  Total, high-density, low-density cholesterol, and triglycerides will be assessed through a blood draws.
Change in body mass index | Baseline, 12 weeks [end of study]
  Height will be measured using a stadiometer to the nearest decimal point in cm. Weight will be measured using a scale to the nearest decimal in kg. Body mass index will be calculated using kg/m^2.
Change in body fat percentage | Baseline, 12 weeks [end of study]
  Body fat percentage will be measured using a scale to the nearest decimal.
Change in waist circumference | Baseline, 12 weeks [end of study]
  Waist circumference will be measured using a waist circumference tape to the nearest decimal in cm.
Change in high blood pressure status | Baseline, 12 weeks [end of study]
  Blood pressure will be measured using blood pressure monitors. High blood pressure is considered as reading of >=120/80.

CONTACTS AND LOCATIONS:
Overall Officials: Tashara M Leak, PhD, RD, Principal Investigator — Cornell University
Locations (1):
- Brownsville Neighborhood Health Action Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No